CLINICAL TRIAL: NCT02858791
Title: MIF- Thyroxine Interactions in the Pathogenesis of Pulmonary Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Arunabh Talwar, Attending Physician, Northwell Health
Other Study IDs: 13-003A
Record Dates: First submitted 2016-06-14; First posted 2016-08-08 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Hypertension; Pulmonary Arterial Hypertension; Interstitial Lung Disease
MeSH Terms: conditions — Hypertension, Pulmonary; Pulmonary Arterial Hypertension; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Venous blood samples will be collected for analysis before and after completing cardiopulmonary exercise test
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Healthy Controls: Subjects are made up of healthy adults
  Interventions:
  Venous blood drawn before and after cardiopulmonary exercise test Will have a resting 12 lead EKG Undergo pulmonary function test
- Affected: Subjects have Pulmonary Hypertension Subjects have Pulmonary hypertension with Interstitial lung disease Subjects have Interstitial lung disease
  Interventions:
  Venous blood drawn before and after cardiopulmonary exercise test Will have a resting 12 lead EKG Undergo pulmonary function test

SUMMARY:
The investigators will investigate the interrelationship of macrophage migration inhibitory factor (MIF) and free T4 in patients with PAH.

DETAILED DESCRIPTION:
The investigators will test our hypothesis and accomplish our objectives by pursuing three Specific Aims:

To investigate the interrelationship between macrophage migration inhibitory factor (MIF) and free T4 in patients with PAH with a working hypothesis that an increased release of MIF into the pulmonary vasculature during cardiopulmonary exercise changes the normal balance between plasma MIF and T4.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be at least 18 years of age and have confirmed pulmonary hypertension (PH) and interstitial lung disease (ILD).
* ILD was identified on high resolution computed tomography along with a total lung capacity (TLC) <70% of predicted value on pulmonary function tests (PFTs) with no evidence of pulmonary hypertension on echocardiogram.
* PAH group patients were defined as patients with a mean pulmonary artery pressure >25 mmHg at rest and a wedge pressure of <15 mmHg (millimeters of mercury), measured by right heart catheterization (WHO group I PAH).
* PH+ILD group, subjects with evidence of ILD on high resolution CT Scan and mean pulmonary artery pressure >25 mmHg on right heart catheterization.
* Patient with evidence of Chronic thromboembolic disease on CT angiogram and mean pulmonary artery pressure >25mmHg on right heart catheterization. (WHO group IV)
* Patient with Pulmonary Hypertension due to other conditions, such as Sarcoidosis, Gauchers disease, Hemolytic Anemia and Myeloproliferative disorders.
* Normal control group: Subjects without cardiopulmonary disease, with a normal PFT and ECG.

Exclusion Criteria:

* Failure to obtain informed consent;
* Pregnancy
* Subjects with cardiopulmonary disease other than PH and ILD;
* Unexplained abnormal PFT, ECG, Routine blood/chemistries test
* History or existing other sever organ/system diseases
* Defined Acute pulmonary embolism
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects are either a healthy volunteer, or patietns who have confirmed pulmonary hypertension and interstitial lung disease
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
To examine the MIF-T4 relationship in patients before/after a standardized exercise challenge | up to 30 mins
  Assess levels of the proinflammatory cytokine macrophage migration inhibitory factor (MIF) before/after standard exercise challenge

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health, New Hyde Park, New York, United States